CLINICAL TRIAL: NCT02415205
Title: Pain and Stress Assessment and ROP Screening Examination in Premature Infants
Brief Title: Pain and Stress Assessment and ROP Screening
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Danilyn Angeles, PhD, PhD, Loma Linda University
Other Study IDs: 5150005
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Pain; Stress
Keywords: Pain and stress assessment in premature infants
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study will measure the effects of eye exams on markers of stress in the urine. In addition, measurements will be taken to show the effects of stress on brain activity, O2 sats, and blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants between 24 -32 weeks of gestational age

Exclusion Criteria:

* Infants scheduled for laser eye surgery on the day of the examination
* Infants with intraventricular hemorrhage ≥ grade 3 (Papile classification) diagnosed by head ultrasound
* Infants receiving the following medications: morphine, fentanyl, methadone, midazolam, lorazepam, muscle relaxants, phenobarbital, phenytoin, levetiracetam
* Renal injury defined with plasma creatinine > 1.5 mg/dL
* Severe cyanotic congenital heart disease
* Unstable respiratory distress (hypoxemia PaO2 < 50 mm Hg or SpO2 < 90%)

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Premature infants undergoing SOC ROP eye exams
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-04; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Urine Stress Marker | 24 hours
  Collection to occur 3-4 hours before eye exam and 24 hours after the eye exam.

SECONDARY OUTCOMES:
aEEG | 24 hours
  1 hour prior to the eye examination and will remain there until 24 hours after the end of the eye exam.
NIRS | 24 hours
  1 hour prior to the eye exam and will be kept in place until 24 hours after the end of the eye exam

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hopper, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Children's Hospital, Loma Linda, California, United States